CLINICAL TRIAL: NCT04978337
Title: A Phase 2b Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Rilematovir (JNJ-53718678) in Adult Outpatients With Respiratory Syncytial Virus (RSV) Infection Who Are at High Risk for RSV-related Disease Progression
Brief Title: A Study of Rilematovir (JNJ-53718678) in Adult Outpatients With Respiratory Syncytial Virus (RSV) Infection
Acronym: PRIMROSE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Janssen made the strategic decision to discontinue the PRIMROSE study. This decision is not based on any safety concerns.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109031; 53718678RSV2008 (Other: Janssen Research & Development, LLC); 2020-005980-30 (EudraCT Number)
Expanded Access: NCT04221412 (No longer available)
Record Dates: First submitted 2021-07-26; First posted 2021-07-27 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Syncytial Virus
MeSH Terms: interventions — JNJ-53718678

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: Rilematovir (Experimental): Participants will receive oral dose of rilematovir 250 milligrams (mg), twice daily (bid) for 7 days.
  Interventions: Drug: Rilematovir
- Treatment B: Placebo (Placebo Comparator): Participants will receive oral dose of placebo matching to rilematovir, bid for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rilematovir — Rilematovir 250 mg will be administered orally.
  Other Names: JNJ-53718678
  Arms: Treatment A: Rilematovir
Drug: Placebo — Placebo matching to rilematovir will be administered orally.
  Arms: Treatment B: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of rilematovir compared to placebo with respect to the time to resolution of respiratory syncytial virus (RSV) lower respiratory tract disease (LRTD) symptoms.

DETAILED DESCRIPTION:
Rilematovir is an investigational RSV specific fusion inhibitor currently in development for the treatment of RSV infection in both adult and pediatric populations. The study will include a Screening period (Day -1 to Day 1), a Treatment period (Day 1 to Day 7/8 [depending on timing of first dose]), and a Follow-up period (Day 8/9 to Day 35). The total study duration of the study for each participant will be up to 35 days. The study will evaluate efficacy and safety of RSV in adult outpatients (18-85 years) who are at high risk of RSV related disease progression and have at least moderate RSV disease. The efficacy assessments include evaluation with electronic patient-reported outcome (ePRO) and the safety assessments include evaluations of physical examinations, vital signs, electrocardiograms, clinical laboratory tests, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Presented to the healthcare facility with symptoms suggestive of a diagnosis of acute respiratory syncytial virus (RSV) infection
* Has at least 2 symptoms of lower respiratory tract disease (LRTD), one of which must be scored as at least 'moderate' if the symptoms did not pre-exist before RSV onset, or one of which is scored worse than usual if the symptoms pre-existed
* Tested positive for RSV infection using a molecular-based diagnostic assay (polymerase chain reaction [PCR] or other) on a bilateral nasal mid-turbinate swab sample
* Has at least one of the following high-risk conditions that predispose them to RSV-related disease progression: a. age greater than or equal to (>=) 65 years, b. congestive heart failure (CHF), c. chronic obstructive pulmonary disease (COPD), d. asthma
* Randomized to study intervention treatment within 72 hours after onset of any of the RSV symptoms or worsening of pre-existing symptoms
* Not be hospitalized during screening (emergency room or hospital observation status for an anticipated duration of less than [<] 24 hours are not considered as hospitalization)

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to rilematovir or to any of the excipients of rilematovir or placebo formulation
* Presence of clinically significant heart arrhythmias, uncontrolled, unstable atrial arrhythmia, or sustained ventricular arrhythmia
* Participant has known or suspected (from medical history or participant examination) chronic or acute hepatitis B or C infection
* Immunocompromised conditions
* Living in institutional care or assisted living facility and also receiving acute care management for any respiratory condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (86):
- United States (35):
  - Central Alabama Research, Birmingham, Alabama
  - Fiel Family and Sports Medicine Clinical Research Advantage, Tempe, Arizona
  - IMD Clinical Trials, Bakersfield, California
  - Hope clinical Research LLC, Canoga Park, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Bensch Clinical Research, LLC, Stockton, California
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - Best Quality Research Inc, Hialeah, Florida
  - Homestead Associates in Research, Inc, Homestead, Florida
  - Care Partners Clinical Research, Jacksonville, Florida
  - Research Institute Of South Florida, Inc., Miami, Florida
  - Pines Care Research Center Inc, Pembroke Pines, Florida
  - Santos Research Center, Tampa, Florida
  - Privia Medical Group, LLC, Fayetteville, Georgia
  - Southcoast Health, Savannah, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - Montana Medical Research, Missoula, Montana
  - Excel Clinical Research, Las Vegas, Nevada
  - Burke Primary Care, Morganton, North Carolina
  - Dayton Clinical Research, Dayton, Ohio
  - Pulmonologist, Critical Care, and Sleep Medicine, Wyomissing, Pennsylvania
  - Piedmont Clinical Research, Fort Mill, South Carolina
  - Texas Health Care, PLLC, Fort Worth, Texas
  - Mercury Clinical Research, Houston, Texas
  - Next Level Urgent Care, Houston, Texas
  - SW Research LLC, Houston, Texas
  - SMS Clinical Research LLC, Mesquite, Texas
  - Rio Grande Valley Clinical Research Institute, Pharr, Texas
  - Javara, San Marcos, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Javara, The Woodlands, Texas
  - CCT Research at South Ogden Family Medicine, South Ogden, Utah
  - Javara, Forest, Virginia
  - Frontier Clinical Research, Morgantown, West Virginia
- Argentina (5):
  - INAER - Investigación en Alergias y Enfermedades Respiratorias, Buenos Aires
  - Centro Respiratorio Quilmes, Quilmes
  - Centro Medico Respire, San Fernando
  - Investigaciones en Patologias Respiratorias, San Miguel de Tucumán
  - Clinica Mayo de UMCB, San Miguel de Tucumán
- Bulgaria (4):
  - Specialized Hospital for Active Treatment of Pneumo-Phthisiatric Diseases-Haskovo Ltd. Haskovo, Haskovo
  - Specialized Hospital for Active Treatment of Pulmonary Diseases - Pernik, Pernik
  - SHAT of Pneumo-phthisiatric Diseases Dr Dimitar Gramatikov - Ruse, EOOD, Rousse
  - Specialized Hospital for Active Treatment of Pulmonary Diseases - Troyan EOOD, Troyan Municipality
- Dr. Anil K Gupta Medicine Professional Corporation, Toronto, Ontario, Canada
- Germany (4):
  - Universitatsklinikum Bonn, Bonn
  - IKF Pneumologie GmbH & Co. KG Am Standort IFS - Interdisziplinäres Facharztzentrum, Frankfurt
  - Gemeinschaftspraxis Dr. Taeschner / Dr. Bonigut, Leipzig
  - Praxis Dr. Weimer, Reinfeld
- Hungary (2):
  - Strázsahegy Medicina Bt, Budapest
  - Omnimodus Elixír Kft., Csorna
- Italy (2):
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Universita Cattolica del Sacro Cuore - Fondazione Policlinico Universitario 'A. Gemelli', Roma
- Japan (7):
  - Nishifukuoka Hospital, Fukuoka
  - Nagata Hospital, Fukuoka
  - Terada Clinic Respiratory Medicine & General Practice, Himeji-shi
  - Kamoike ENT allergy clinic, Kagoshima
  - Shinkomonji hospital, Kitakyushu
  - Koyama Medical Clinic, Nagano
  - Tokyo Shinagawa Hospital, Shinagawa-ku
- Poland (5):
  - Gabinet Lekarski Pediatryczno-Alergologiczny, Bialystok
  - NZOZ Poradnie Specjalistyczne ATOPIA, Krakow
  - ETG Lodz, Lodz
  - Centrum Innowacyjnych Terapii Sp. z o.o., Piaseczno
  - Centrum Badan Klinicznych, Osrodek Badan Wczesnej Fazy, Wroclaw
- South Africa (2):
  - Clinical Trial Systems (Pty) Ltd, Gauteng
  - Private Practice - Dr. Peter Sebastian, KwaZulu-Natal
- Spain (6):
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp. Quiron Barcelona, Barcelona
  - Hosp. Gral. Univ. de Elche, Elche
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Virgen Macarena, Seville
  - Hosp. Clinico Univ. De Valencia, Valencia
- Sweden (4):
  - Skanes universitetssjukhus, Malmo
  - PharmaSite, Malmo
  - ClinSmart Sweden AB, Solna
  - Akademiska Sjukhuset, Uppsala
- Thailand (3):
  - The Hospital for Tropical Diseases, Bangkok
  - Bamrasnaradura Infectious Disease Institute, Nonthaburi
  - King Chulalongkorn Memorial Hospital, Pathumwan
- Ukraine (6):
  - Medical Unit Of Company 'Kharkiv Tractor Plant', Kharkiv Medical Academy Of Postgraduate Education, Kharkiv
  - City Clinical Hospital #1, Kyiv
  - Kyiv Railway Clinical Hospital #2 Of Branch 'Health Center' Of The Company 'Ukrainian Railway', Kyiv
  - Medical Center 'Consylium Medical', Kyiv
  - Policlinic of State Joint Stock Holding Company 'Artem', Kyiv
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participant received oral dose of placebo matching to rilematovir twice daily for 7 days.
- Rilematovir 250 mg Bid: Participants received oral dose of rilematovir 250 milligrams (mg) twice daily for 7 days.
Period: Overall Study
Arm/Group | Placebo | Rilematovir 250 mg Bid
Started | 1 | 4
Completed | 1 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rilematovir 250 mg Bid | Total
Number analyzed (Participants) | 1 | 4 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 | 51.8 (22.9) | 52.4 (19.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 4 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  BULGARIA | 1 | 0 | 1
  HUNGARY | 0 | 1 | 1
  POLAND | 0 | 1 | 1
  UNITED STATES | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Syncytial Virus (RSV) Lower Respiratory Tract Disease (LRTD) Symptoms as Assessed by Respiratory Infection Intensity and Impact Questionnaire (RiiQ) Symptom Scale Score at Baseline
Description: RSV LRTD symptoms (cough, short of breath, wheezing, coughing up phlegm [sputum]) as assessed by the RiiQ symptom scale score at baseline were reported. The RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The LRTD symptom score was calculated as the mean of the LRTD symptom scores.
Time Frame: Baseline
Population: Intent-to-Treat infected (ITT-i) analysis set included all participants who were randomized and treated (at least one dose) and had RSV infection confirmed by central laboratory analysis. Participants with confirmed severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) infection (positive test by central laboratory analysis) were excluded.
Measure: Number; unit: Scores on a scale
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 4
Scores on a scale
  Participant 1: number analyzed (Participants) | 0 | 1
  Participant 1 |  | 1.25
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 1.25
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 1.25
  Participant 4: number analyzed (Participants) | 0 | 1
  Participant 4 |  | 2.25
  Participants 5: number analyzed (Participants) | 1 | 0
  Participants 5 | 2.25 |

2. Secondary Outcome: Percentage of Participants With Post-Baseline RSV-related Complications
Description: RSV-related complications were reported. The RSV-related complications included pulmonary complications (primary viral pneumonia, bronchitis, respiratory failure, secondary bacterial pneumonia, and exacerbations of underlying chronic pulmonary diseases [such as COPD and asthma]) and extrapulmonary complications (cardiovascular and cerebrovascular disease events, congestive heart failure [CHF] or exacerbation of underlying CHF, acute exacerbation of chronic kidney disease, severe dehydration, decompensation of previously controlled diabetes mellitus, and other airway infections). Complications after first intake of study drug were considered for this outcome measure.
Time Frame: Up to Day 35
Population: ITT-i analysis set included all participants who were randomized and treated (at least one dose) and had RSV infection confirmed by central laboratory analysis. Participants with confirmed SARS-CoV-2 infection (positive test by central laboratory analysis) were excluded.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 4
Percentage of participants | 0 | 0

3. Secondary Outcome: Percentage of Participants With New Antibiotic Use, or New Use or Increased Dose of Systemic or Inhaled Corticosteroids and Bronchodilator, or Home Oxygen Supplementation
Description: New antibiotic use, or new use or increased dose of systemic or inhaled corticosteroids and bronchodilators, or home oxygen supplementation were reported.
Time Frame: Up to Day 35
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 4
Percentage of participants
  New antibiotic use | 0 | 25.0
  New use or increased dose of systematic or inhaled corticosteroids and bronchodilators | 0 | 25.0
  Home oxygen supplementation | 0 | 0

4. Secondary Outcome: Percentage of Participants With Unscheduled Outpatient Clinic Visits, Emergency Room Visits or Hospitalization for Respiratory Infection
Description: Unscheduled outpatient clinic visits, emergency room visits or hospitalization for respiratory infection were reported.
Time Frame: Up to Day 35
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 4
Percentage of participants
  Unscheduled outpatient clinic visits | 0 | 25.0
  Emergency room visits | 0 | 0
  Hospitalization for respiratory infection | 0 | 0

5. Secondary Outcome: Percentage of Participants Meeting a Composite Endpoint of Either Developing RSV-Related Complications and/or Needing RSV-related Medical Attendance
Description: Percentage of participants meeting a composite endpoint of either developing RSV-related complications (pulmonary and extra-pulmonary) and/or needing RSV-related medical attendance was derived.
Time Frame: Up to Day 35
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 4
Percentage of participants | 0 | 25.0

6. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse events (AEs) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Any AE which occurred at or after the initial administration of study intervention through the end of the study (that is, Day 35) was considered treatment-emergent.
Time Frame: Up to Day 35
Population: Safety analysis set included all participants who took at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 4
Percentage of participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With Treatment-emergent Abnormal Clinical Laboratory Findings
Description: Abnormal clinical laboratory findings were reported. Laboratory abnormalities were determined as per division of microbiology and infectious diseases(DMID) toxicity as Grade 1:mild(transient or mild discomfort [less than {<} 48 hours]; no medical intervention/therapy required); Grade 2:moderate (mild to moderate limitation in activity-some assistance may be needed; no or minimal medical intervention/therapy required); Grade 3:severe (severe marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible); Grade 4:life-threatening (extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable). Only Grade 2 abnormalities are reported in this outcome measure. A treatment emergent abnormality is any abnormality not present at baseline and occurring post first administration or worsening versus baseline post first administration.
Time Frame: Up to Day 35
Population: Safety analysis set included all participants who took at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 4
Percentage of participants
  Decrease in hemoglobin (Grade 2) | 0 | 25
  Increase in glucose (Grade 2) | 0 | 25

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Abnormalities in Electrocardiograms (ECGs)
Description: Various ECG variables assessed were heart rate: abnormally low (less than or equal to [<=] 45 beats per minute [bpm]), abnormally high (greater than or equal to [>=] 120 bpm); PR interval: abnormally high (>=210 milliseconds [msec]); QRS interval: abnormally high (>=120 msec); QTc: borderline prolonged: >450 msec and <=480 msec, prolonged: >480 msec and <=500 msec, pathologicaly prolonged: >500 msec. A treatment emergent abnormality is any abnormality not present at baseline and occurring post first administration or worsening versus baseline post first administration.
Time Frame: Up to Day 35
Population: Safety analysis set included all participants who took at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 4
Percentage of participants | 0 | 0

9. Secondary Outcome: Percentage of Participants With Treatment-emergent Abnormal Vital Signs Findings
Description: Abnormal vital parameters included pulse rate: abnormally low <=45 bpm, abnormally high >=120 bpm; Systolic Blood Pressure (SBP): abnormally low <=90 millimeter of mercury (mmHg), Grade 1 (mild): >140 mmHg to <160 mmHg, Grade 2 (moderate): >=160 mmHg to <180 mmHg, Grade 3 (severe): >=180 mmHg; Diastolic BP: abnormally low <=50 mmHg, Grade 1: >90 mmHg to <100 mmHg, Grade 2: >=100 mmHg to <110 mmHg, Grade 3: >=110 mmHg; Respiratory rate: Grade 1 (mild): 17-20 breaths per minute, Grade 2 (moderate): 21-25 breaths per minute, Grade 3 (severe): >25 breaths per minute, Grade 4 (potentially life threatening): intubation; Oxygen saturation: abnormally low: <95%; Temperature: abnormally high >38.0 degree celsius. A treatment emergent abnormality is any abnormality not present at baseline and occurring post first administration or worsening versus baseline post first administration.
Time Frame: Up to Day 35
Population: Safety analysis set included all participants who took at least 1 dose of study intervention.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 4
Percentage of participants | 0 | 0

10. Secondary Outcome: RSV Viral Load Over Time
Description: RSV viral load (subtype: RSV A and RSV B) was measured over time by quantitative reverse transcription polymerase chain reaction (qRT-PCR) in the nasal swab specimens collected at the clinic visits and at home. In this outcome measure, only those timepoints and RSV subtypes (A or B) for which individual participants had data were reported.
Time Frame: Baseline, Days 3, 5, 8, 15, and 21
Population: ITT-i analysis set included all participants who were randomized and treated (at least one dose) and had RSV infection confirmed by central laboratory analysis. Participants with confirmed SARS-CoV-2 infection (positive test by central laboratory analysis) were excluded. Here, 'N' (number of participants analyzed) signifies number of participants with available data for this outcome measure and 'n' (number analyzed) represents number of participants evaluable at the specified timepoints.
Measure: Number; unit: log10 copies per milliliter (mL)
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 3
log10 copies per milliliter (mL)
  Participant 1: Baseline: RSV B: number analyzed (Participants) | 0 | 1
  Participant 1: Baseline: RSV B |  | 6.87
  Participant 1: Day 3: RSV B: number analyzed (Participants) | 0 | 1
  Participant 1: Day 3: RSV B |  | 5.84
  Participant 1: Day 8: RSV B: number analyzed (Participants) | 0 | 1
  Participant 1: Day 8: RSV B |  | 0
  Participant 1: Day 15: RSV B: number analyzed (Participants) | 0 | 1
  Participant 1: Day 15: RSV B |  | 0
  Participant 1: Day 21: RSV B: number analyzed (Participants) | 0 | 1
  Participant 1: Day 21: RSV B |  | 0
  Participant 2: Baseline: RSV B: number analyzed (Participants) | 0 | 1
  Participant 2: Baseline: RSV B |  | 6.17
  Participant 2: Day 3: RSV B: number analyzed (Participants) | 0 | 1
  Participant 2: Day 3: RSV B |  | 6.71
  Participant 2: Day 8: RSV B: number analyzed (Participants) | 0 | 1
  Participant 2: Day 8: RSV B |  | 0
  Participant 2: Day 15: RSV B: number analyzed (Participants) | 0 | 1
  Participant 2: Day 15: RSV B |  | 0
  Participant 2: Day 21: RSV B: number analyzed (Participants) | 0 | 1
  Participant 2: Day 21: RSV B |  | 0
  Participant 3: Baseline: RSV A: number analyzed (Participants) | 0 | 1
  Participant 3: Baseline: RSV A |  | 6.5
  Participant 3: Day 3: RSV A: number analyzed (Participants) | 0 | 1
  Participant 3: Day 3: RSV A |  | 6.4
  Participant 3: Day 5: RSV A: number analyzed (Participants) | 0 | 1
  Participant 3: Day 5: RSV A |  | 3.37
  Participant 3: Day 8: RSV A: number analyzed (Participants) | 0 | 1
  Participant 3: Day 8: RSV A |  | 2.9
  Participant 3: Day 15: RSV A: number analyzed (Participants) | 0 | 1
  Participant 3: Day 15: RSV A |  | 0
  Participant 3: Day 21: RSV A: number analyzed (Participants) | 0 | 1
  Participant 3: Day 21: RSV A |  | 0
  Participant 5: Baseline: RSV A: number analyzed (Participants) | 1 | 0
  Participant 5: Baseline: RSV A | 7.57 |
  Participant 5: Day 3: RSV A: number analyzed (Participants) | 1 | 0
  Participant 5: Day 3: RSV A | 4.94 |
  Participant 5: Day 5: RSV A: number analyzed (Participants) | 1 | 0
  Participant 5: Day 5: RSV A | 0 |
  Participant 5: Day 8: RSV A: number analyzed (Participants) | 1 | 0
  Participant 5: Day 8: RSV A | 0 |
  Participant 5: Day 15: RSV A: number analyzed (Participants) | 1 | 0
  Participant 5: Day 15: RSV A | 0 |
  Participant 5: Day 21: RSV A: number analyzed (Participants) | 1 | 0
  Participant 5: Day 21: RSV A | 0 |

11. Secondary Outcome: Plasma Concentration of Rilematovir
Description: Plasma concentration of rilematovir was reported. This outcome measure was planned to be analyzed for specified arm only. In this outcome measure, only those timepoints for which individual participants had data were reported.
Time Frame: Day 1: 1 hour post dose, Day 3: pre-dose and 1 hour post dose, and Follow-up: Day 8
Population: Pharmacokinetic (PK) analysis set included all participants who were randomized and treated (at least one dose) and had RSV infection confirmed by central laboratory analysis. Here, 'N' (number of participants analyzed) signifies number of participants with available data for this outcome measure.
Measure: Number; unit: Nanograms per milliliter (ng/mL)
Arm/Group | Rilematovir 250 mg Bid
Number analyzed (Participants) | 3
Nanograms per milliliter (ng/mL)
  Participant 1: Day 3 (Pre-dose): number analyzed (Participants) | 1
  Participant 1: Day 3 (Pre-dose) | 658
  Participant 1: Day 3 (1 hour post dose): number analyzed (Participants) | 1
  Participant 1: Day 3 (1 hour post dose) | 682
  Participant 1: Follow-up-Day 8: number analyzed (Participants) | 1
  Participant 1: Follow-up-Day 8 | 9.63
  Participant 2: Day 3 (pre-dose): number analyzed (Participants) | 1
  Participant 2: Day 3 (pre-dose) | 15.9
  Participant 2: Day 3 (1 hour post dose): number analyzed (Participants) | 1
  Participant 2: Day 3 (1 hour post dose) | 465
  Participant 2: Follow-up-Day 8: number analyzed (Participants) | 1
  Participant 2: Follow-up-Day 8 | 494
  Participant 3: Day 1 (1 hour post dose): number analyzed (Participants) | 1
  Participant 3: Day 1 (1 hour post dose) | 257
  Participant 3: Day 3 (pre-dose): number analyzed (Participants) | 1
  Participant 3: Day 3 (pre-dose) | 2400
  Participant 3: Day 3 (1 hour post dose): number analyzed (Participants) | 1
  Participant 3: Day 3 (1 hour post dose) | 2960
  Participant 3: Follow-up-Day 8: number analyzed (Participants) | 1
  Participant 3: Follow-up-Day 8 | 3130

12. Primary Outcome: Respiratory Syncytial Virus (RSV) Lower Respiratory Tract Disease (LRTD) Symptoms as Assessed by Respiratory Infection Intensity and Impact Questionnaire (RiiQ) Symptom Scale Score at Day 3
Description: RSV LRTD symptoms (cough, short of breath, wheezing, coughing up phlegm [sputum]) as assessed by the RiiQ symptom scale score at Day 3 were reported. The RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The LRTD symptom score was calculated as the mean of the LRTD symptom scores. In this outcome measure, only those individual participants who had data were reported.
Time Frame: Day 3
Population: ITT-I analysis set included all participants who were randomized and treated (at least one dose) and had RSV infection confirmed by central laboratory analysis. Participants with confirmed SARS-CoV-2 infection (positive test by central laboratory analysis) were excluded. Here, 'N' (number of participants analyzed) signifies number of participants with available data for this outcome measure.
Measure: Number; unit: Scores on a scale
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 1
Scores on a scale
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 0.75
  Participant 5: number analyzed (Participants) | 1 | 0
  Participant 5 | 1.75 |

13. Primary Outcome: Respiratory Syncytial Virus (RSV) Lower Respiratory Tract Disease (LRTD) Symptoms as Assessed by Respiratory Infection Intensity and Impact Questionnaire (RiiQ) Symptom Scale Score at Day 8
Description: RSV LRTD symptoms (cough, short of breath, wheezing, coughing up phlegm [sputum]) as assessed by the RiiQ symptom scale score at Day 8 were reported. The RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The LRTD symptom score was calculated as the mean of the LRTD symptom scores. In this outcome measure, only those individual participants who had data were reported.
Time Frame: Day 8
Population: as for outcome 12
Measure: Number; unit: Scores on a scale
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 3
Scores on a scale
  Participant 1: number analyzed (Participants) | 0 | 1
  Participant 1 |  | 1.25
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 1.25
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 0.75
  Participant 5: number analyzed (Participants) | 1 | 0
  Participant 5 | 0.5 |

14. Primary Outcome: Respiratory Syncytial Virus (RSV) Lower Respiratory Tract Disease (LRTD) Symptoms as Assessed by Respiratory Infection Intensity and Impact Questionnaire (RiiQ) Symptom Scale Score at Day 14
Description: RSV LRTD symptoms (cough, short of breath, wheezing, coughing up phlegm [sputum]) as assessed by the RiiQ symptom scale score at Day 14 were reported. The RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The LRTD symptom score was calculated as the mean of the LRTD symptom scores. In this outcome measure, only those individual participants who had data were reported.
Time Frame: Day 14
Population: as for outcome 12
Measure: Number; unit: Scores on a scale
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 3
Scores on a scale
  Participant 1: number analyzed (Participants) | 0 | 1
  Participant 1 |  | 1.25
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 1
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 0
  Participant 5: number analyzed (Participants) | 1 | 0
  Participant 5 | 0 |

15. Primary Outcome: Respiratory Syncytial Virus (RSV) Lower Respiratory Tract Disease (LRTD) Symptoms as Assessed by Respiratory Infection Intensity and Impact Questionnaire (RiiQ) Symptom Scale Score at Day 21
Description: RSV LRTD symptoms (cough, short of breath, wheezing, coughing up phlegm [sputum]) as assessed by the RiiQ symptom scale score at Day 21 were reported. The RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The LRTD symptom score was calculated as the mean of the LRTD symptom scores. In this outcome measure, only those individual participants who had data were reported.
Time Frame: Day 21
Population: as for outcome 12
Measure: Number; unit: Scores on a scale
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 3
Scores on a scale
  Participant 1: number analyzed (Participants) | 0 | 1
  Participant 1 |  | 0
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 1
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 0
  Participant 5: number analyzed (Participants) | 1 | 0
  Participant 5 | 0 |

16. Primary Outcome: Respiratory Syncytial Virus (RSV) Lower Respiratory Tract Disease (LRTD) Symptoms as Assessed by Respiratory Infection Intensity and Impact Questionnaire (RiiQ) Symptom Scale Score at Day 28
Description: RSV LRTD symptoms (cough, short of breath, wheezing, coughing up phlegm [sputum]) as assessed by the RiiQ symptom scale score at Day 28 were reported. The RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The LRTD symptom score was calculated as the mean of the LRTD symptom scores. In this outcome measure, only those individual participants who had data were reported.
Time Frame: Day 28
Population: as for outcome 12
Measure: Number; unit: Scores on a scale
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 3
Scores on a scale
  Participant 1: number analyzed (Participants) | 0 | 1
  Participant 1 |  | 0.5
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 0.75
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 0
  Participant 5: number analyzed (Participants) | 1 | 0
  Participant 5 | 0 |

17. Primary Outcome: Respiratory Syncytial Virus (RSV) Lower Respiratory Tract Disease (LRTD) Symptoms as Assessed by Respiratory Infection Intensity and Impact Questionnaire (RiiQ) Symptom Scale Score at Day 35
Description: RSV LRTD symptoms (cough, short of breath, wheezing, coughing up phlegm [sputum]) as assessed by the RiiQ symptom scale score at Day 35 were reported. The RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The LRTD symptom score was calculated as the mean of the LRTD symptom scores. In this outcome measure, only those individual participants who had data were reported.
Time Frame: Day 35
Population: as for outcome 12
Measure: Number; unit: Scores on a scale
Arm/Group | Placebo | Rilematovir 250 mg Bid
Number analyzed (Participants) | 1 | 3
Scores on a scale
  Participant 1: number analyzed (Participants) | 0 | 1
  Participant 1 |  | 0
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 0
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 0
  Participant 5: number analyzed (Participants) | 1 | 0
  Participant 5 | 0 |

ADVERSE EVENTS:
Time Frame: Up to Day 35
Description: Safety analysis set included all participants who took at least 1 dose of study intervention.
Arm/Group | Placebo | Rilematovir 250 mg Bid
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 0/4

LIMITATIONS AND CAVEATS:
As the study was terminated early, a low number of participants were enrolled, hence some efficacy analyses were not performed per change in the planned analysis. Thereby, data were analyzed for safety and selected efficacy parameters only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will with hold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04978337/Prot_002.pdf
  • Statistical Analysis Plan (2022-05-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT04978337/SAP_003.pdf